CLINICAL TRIAL: NCT06046365
Title: Early Diagnosis of Breast Cancer-related Lymphedema
Status: Recruiting | Type: Observational
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Zheng-Yu Hoe, MD., PhD., Chairperson, Kaohsiung Veterans General Hospital.
Other Study IDs: 22-CT2-15(211230-3)
Record Dates: First submitted 2023-08-28; First posted 2023-09-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Lymphedema
Keywords: lymphoedema; limb circumference; tissue hardness
MeSH Terms: conditions — Lymphedema | interventions — Lymphoscintigraphy; Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- mastectomy: Expected to include female patients who are undergoing breast cancer resection surgery or those who have already undergone breast resection surgery for breast cancer.
  Interventions: Diagnostic Test: lymphoscintigraphy; Diagnostic Test: circumference measurement; Diagnostic Test: sonography; Diagnostic Test: DXA body composition analysis

INTERVENTIONS:
Diagnostic Test: lymphoscintigraphy — lymphoscintigraphy
Diagnostic Test: circumference measurement — circumference measurement
Diagnostic Test: sonography — B-mode sono and elastography
Diagnostic Test: DXA body composition analysis — DXA body composition analysis

SUMMARY:
This study will conduct clinical trials to explore the mechanisms behind the development of upper limb lymphedema following breast cancer surgery. The investigators will recruit patients who have undergone breast cancer surgery and utilize Indocyanine Green (ICG) lymphography and Lymphoscintigraphy to identify the locations of lymphatic blockages. Shear Wave Elastography (SWE) will be used to detect changes in tissue limb compliance. DXA body composition analysis will measure the differences in the composition ratios between edematous and normal limbs. In addition, diffusion correlation spectrometry will be employed to monitor changes in deep tissue blood flow, complemented by continuous measurements of limb circumference and other physiological parameters. The study aims to explore the interrelationships among lymphatic circulation, limb circumference, tissue compliance, and tissue blood flow rates.

DETAILED DESCRIPTION:
Breast cancer ranks as the most common cancer among women in Taiwan. According to the cancer registry data of Taiwan's Ministry of Health and Welfare, there were 16,325 new cases of breast cancer in 2016. Approximately one in 12 women will develop breast cancer in her lifetime. Although the incidence rate is high, the survival rate after clinical treatment is also quite high. The five-year survival rate for early-stage breast cancer patients exceeds 90%, making it a highly manageable disease at present.

The incidence rate of breast cancer-related lymphedema is around 21.4%, and is expected to become increasingly common as the survival rate of patients improves. Aside from causing psychological distress, it also impairs a patient's work and daily life capabilities. Patients also have to bear additional medical expenses, which brings a significant financial burden to families. Current research supports that early detection and treatment are key to controlling breast cancer-related lymphedema. However, there is still a need for a clearer understanding of the risk factors causing lymphedema and the physiological changes that occur when it manifests, in order to achieve the goal of early detection.

This study will conduct clinical trials to investigate the mechanisms of upper limb lymphedema after breast cancer surgery. The investigators will recruit post-operative breast cancer patients and use Indocyanine Green (ICG) lymphography and Lymphoscintigraphy to detect lymphatic blockage locations; Shear Wave Elastography (SWE) to detect changes in tissue limb compliance; DXA body composition analysis to measure the differences in edema and normal limb composition ratios; and diffusion correlation spectrometry to measure deep tissue blood flow changes, along with continuous measurements of limb circumference and other physiological parameters. The study aims to explore the interrelationship among lymphatic circulation, limb circumference, tissue compliance, and tissue blood flow.

The expected results of this study can help the investigators understand the risk factors causing lymphedema and the physiological changes that occur when it manifests, overcome the current difficulties in early lymphedema detection, and develop effective monitoring methods and equipment. This will provide more possibilities for the early detection and treatment of future patients with breast cancer-related lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who are expected to undergo breast cancer resection surgery or have already undergone breast resection surgery for breast cancer.
* Absence of unhealed open wounds or other conditions unsuitable for tactile measurements within the measurement area.
* No severe cognitive or emotional impairments.
* No substance abuse (alcohol or drugs).
* Females aged between 20 and 80, capable of fully complying with the requirements of this study plan.

Exclusion Criteria:

* Presence of unhealed open wounds or other conditions unsuitable for tactile measurements within the measurement area.
* Upper limb abnormalities in function (including joint mobility and muscle strength).
* Significant cognitive, auditory, or expressive language issues that hinder comprehension and compliance with instructions.
* Lack of assistance for daily measurements.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aims to recruit 100 breast cancer patients (those who have previously undergone or are expected to undergo any form of breast resection surgery) for research purposes.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
circumference | everyday, through study completion, an average of 1 year
  Circumference measurements are taken and recorded at 2 cm intervals from the wrist crease to the armpit on both upper limbs
Tissue compliance | every 1 week, through study completion, an average of 1 year
  Measurements are taken every 5 cm from the wrist crease to the armpit on both upper limbs using ShearWave Elastography
Lymphoscintigraphy | Once at the beginning of the study, and another assessment will be conducted six months later if there is a deterioration in lymphedema
  Golden Standard for diagnosing lymphedema, used for detecting the location of lymphatic circulation blockage
Indocyanine green (ICG) lymphography | Once at the beginning of the study, and another assessment will be conducted 3 months later if there is a deterioration in lymphedema
  Routine examination, used for detecting the type of lymphatic blockage
DXA body composition analysis | Once at the beginning of the study, and another assessment will be conducted 3 months later if there is a deterioration in lymphedema
  Using DXA to detect and compare the composition of both limbs at different stages after the onset of lymphedema, including changes in protein, fat, and mineral density

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available